CLINICAL TRIAL: NCT04530812
Title: Pilot Study of Fermented Milk Supplementation on Symptoms of Disease and Treatment in Patients With Multiple Myeloma
Brief Title: Fermented Milk Supplementation on Symptoms of Disease and Treatment in Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 657720; NCI-2020-05777 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 657720 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Practice Guidelines as Topic; Standard of Care; Kefir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (commercial kefir beverage) (Experimental): Patients consume commercial kefir beverage daily for 3 months.
  Interventions: Dietary Supplement: Kefir; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual diet) (Active Comparator): Patients maintain usual diet for 3 months.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Maintain usual diet
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual diet)
Dietary Supplement: Kefir — Consume commercial kefir beverage
  Other Names: Kephir
  Arms: Arm I (commercial kefir beverage)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial investigates the effect of fermented milk supplementation on symptoms of disease and treatment in patients with multiple myeloma. Patients with multiple myeloma may experience symptoms related to the disease and/or treatment that affect quality of life. Supplementing usual diet with a probiotic fermented milk product called kefir may contribute to reducing disease and treatment-related side effects through changing the intestinal bacteria community structure and related metabolism.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of a 3-month randomized dietary intervention with a probiotic kefir beverage in multiple myeloma (MM) patients on biomarkers of metabolism, and patient-reported pain and fatigue, gut health, and quality of life (QoL).

SECONDARY OBJECTIVE:

I. Determine the effect of kefir supplementation on gut microbial phylotype and predicted bacterial metabolic function, and assess associations with biomarkers of metabolism, and patient-reported pain and fatigue, gut health, and QoL.

EXPLORATORY OBJECTIVE:

I. Feasibility of a probiotic lifestyle intervention in MM patients.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients consume commercial kefir beverage daily for 3 months.

ARM II: Patients maintain usual diet for 3 months.

After completion of study, patients are followed up at 30 days or until resolution of any study related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Neutrophil values > 1,000/uL
* Diagnosis of multiple myeloma: on maintenance or continued treatment
* Show no signs of comorbidities, myeloma symptoms, or treatment side effects that would put them in danger when participating in the study according to the physician's discretion
* Able to understand and comply with study instructions, including willing to purchase and consume study beverage daily if in intervention arm or, avoid regular consumption of fermented dairy foods (kefir, yogurt, lassi, etc.) if in the control arm
* Understand the investigational nature of the study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Allergies to milk
* Lactose intolerance
* Current habitual (> 3 times per week) consumption of yogurt, kefir, lassi, over-the-counter probiotic dietary supplements
* Chronic inflammatory bowel disease
* Autologous stem cell transplantation or chimeric antigen receptor (CAR)-T cell therapy within the last 6 months
* Prior allogeneic stem cell transplantation
* Major comorbidities that would cause danger to the patient when participating in the study
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to take part in study intervention
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in levels of parathyroid hormone (PTH) | Week 12
  Collect Changes in values of PTH from baseline to week 12in patients who added kefir to their diet
Change in quality of life | Up to 30 days post-intervention
  Will be assessed by European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life-Core 30 and EORTC Myeloma module. Will compare the changes in outcomes pre- to post-intervention between groups using an ANCOVA model

SECONDARY OUTCOMES:
Overall Gut microbial community structure | At baseline and after 3 months daily kefir consumption
  Will evaluate changes in microbial community structure, measured as a beta diversity metric. These changes will be assessed using a regression based kernel association test. Unrarefied phyla, genera, species, and imputed functional genes in pathways will be center log ratio transformed to better approximate a normal distribution. Linear mixed models adjusting for sex, age, body fat mass, energy intake, and baseline measures will be used to evaluate differences in response between diets for alpha diversity, individual phyla, genera, species, and imputed functional gene pathways.

OTHER OUTCOMES:
Symptom Improvement | Up to 30 days post-intervention
  Feasibility of a probiotic lifestyle intervention in multiple myeloma patients

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States